CLINICAL TRIAL: NCT02520128
Title: A Phase II Study of Intensity Modulated Radiotherapy (IMRT) for Patients With Primary Bone and Soft Tissue Sarcoma
Brief Title: A Study of IMRT in Primary Bone and Soft Tissue Sarcoma
Acronym: IMRiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); NCRI Radiotherapy Trials QA (RTTQA) Group (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/13/0376; C2921/A17558 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2015-07-31; First posted 2015-08-11 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Soft Tissue Sarcoma, Adult; Ewing Sarcoma; Bone Sarcoma; Chordoma
Keywords: Intensity Modulated Radiotherapy; Radiotherapy
MeSH Terms: conditions — Sarcoma; Sarcoma, Ewing; Bone Neoplasms; Chordoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (closed to recruitment) (Other): Cohort 1: Patients with Limb/limb girdle soft tissue sarcoma (STS) receiving (neo)-adjuvant radiotherapy (Intensity Modulated Radiotherapy)
  Dose schedules for Cohort 1:
  * Pre-operative RT - 50 Gy in 25 daily fractions over 5 weeks
  * Post-operative RT - 60 Gy in 30 daily fractions to the high dose planning target volume (PTV) and 52.2 Gy in 30 daily fractions to the low dose PTV treated concurrently over 6 weeks
  * Post-operative RT (positive resection margins) - 66 Gy in 33 daily fractions to the high dose PTV, and 53.46Gy in 33 fractions to the low dose PTV treated concurrently over 6 ½ weeks.
  Interventions: Radiation: Intensity modulated radiotherapy (IMRT)
- Cohort 2 (Other): Cohort 2: Patients with Ewing sarcoma of the spine/pelvis receiving definitive radical or (neo)-adjuvant radiotherapy (Intensity Modulated Radiotherapy)
  Dose schedules for Cohort 2:
  * Pre-operative RT - 50.4 Gy in 28 daily fractions over 5½ weeks
  * Post-operative RT - 54 Gy in 30 daily fractions over 6 weeks
  * Primary RT - 54 Gy in 30 daily fractions over 6 weeks.
  Interventions: Radiation: Intensity modulated radiotherapy (IMRT)
- Cohort 3 (Other): Cohort 3: Patients with non-Ewing primary bone sarcomas of the spine/pelvis receiving definitive radical or adjuvant Radiotherapy (Intensity Modulated Radiotherapy)
  Dose schedule for Cohort 3:
  * Primary RT - 70 Gy in 35 daily fractions over 7 week
  * Post-operative RT (non-chordoma) - primary bone sarcoma 60 Gy in 30 daily fractions over 6 weeks
  * Post-operative RT (chordoma) - 70 Gy in 35 daily fractions over 7 weeks.
  Interventions: Radiation: Intensity modulated radiotherapy (IMRT)

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy (IMRT) — Intensity modulated radiotherapy (IMRT) is an advanced radiotherapy technique that is able to deliver a highly conformal dose to a target with improved sparing of the surrounding normal tissues from moderate to high radiation doses. IMRT is likely to be of particular benefit for tumours that have complex shapes, or those in close proximity to sensitive normal tissues and critical organs. Reducing the dose to normal tissues may in turn reduce the acute and late side effects of treatment. IMRT can be delivered from multiple fixed beam angles or through rotational arc applications such as volumetric modulated arc therapy (VMAT) and tomotherapy. The radiotherapy is delivered using multiple small beams (beamlets) of non-uniform intensity.

SUMMARY:
IMRiS is a phase II trial which aims to assess the feasibility, efficacy and toxicity of Intensity Modulated Radiotherapy (IMRT) in three different cohorts of patients with primary bone and soft tissue sarcoma and to demonstrate whether IMRT can improve on current clinical outcomes.

Cohort 1 of the trial is now closed to recruitment.

DETAILED DESCRIPTION:
IMRiS is a prospective multicentre phase II trial of Intensity Modulated Radiotherapy (IMRT). The trial is aiming to evaluate the role of intensity modulated radiotherapy (IMRT) in soft tissue and bone sarcomas. Three separate sarcoma cohorts will be studied and will be analysed separately. Patients will be enrolled in one of three cohorts depending on the type of sarcoma they have:

Cohort 1- Patients with Limb/limb girdle soft tissue sarcoma receiving (neo)-adjuvant radiotherapy. (closed to recruitment)

Cohort 2- Patients with Ewing sarcoma of the spine/pelvis receiving definitive radical or (neo)-adjuvant radiotherapy.

Cohort 3- Patients with non-Ewing primary bone sarcomas of the spine/pelvis receiving definitive radical or adjuvant radiotherapy.

Dose schedules for each Cohort have been indicated in the Trial Arm description.

Radiotherapy will be delivered with fixed beam IMRT, arc IMRT techniques, or tomotherapy. All trial patients will be followed up until death or a maximum of three years from the date of registration in the trial.

The theoretical advantage to IMRT is the potential reduction in late toxicity and subsequent potential for functional improvement. There have been no prospective studies to date powered to address this, particularly where IMRT is used post-operatively. IMRiS cohort 1 will address this question and establish if the use of IMRT will reduce late normal tissue toxicity.

In cohorts 2 & 3, the aim is to establish if the use of IMRT will enable the achievement of a radiotherapy treatment plan that delivers the optimal dose while keeping within normal tissue tolerances. There have been no clinical trials of IMRT in Ewing sarcoma and there is very little published on the use of IMRT in high grade bone sarcomas and chordomas. It is important to establish the feasibility of IMRT to achieve the required radiation doses to the tumour, and to prospectively document the side effects of treatment in this setting. IMRiS will address this in cohort 2 and cohort 3.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven soft tissue sarcoma of the upper or lower limb or limb girdle (Cohort 1), OR,

   Ewing sarcoma of bone arising in the pelvis or spine (Cohort 2) , OR,

   High grade primary bone sarcoma (non-Ewing) or Chordoma arising in the pelvis/spine (Cohort 3)
2. Patients requiring (neo)adjuvant or definitive radical radiotherapy
3. WHO performance status 0-2
4. Patients aged 16 years or more
5. Patients fit enough to undergo radiotherapy treatment and willing to attend follow up visits as per protocol
6. Women of child-bearing potential must have a negative pregnancy test prior to trial entry. Female patients of child-bearing potential and male patients with partners of child-bearing potential must agree to use adequate contraception methods, which must be continued for 3 months after completion of treatment.
7. Capable of giving written informed consent

Exclusion Criteria:

1. Previous radiotherapy to the same site
2. Patients receiving concurrent chemotherapy with radiotherapy (neo-adjuvant chemotherapy prior to radiotherapy is permitted.
3. Patient with bone sarcomas eligible for proton beam radiotherapy; N.B. if a patient is not to have PBRT for whatever reason, they may be considered for IMRiS.
4. Paediatric type alveolar or embryonal rhabdomyosarcomas
5. Pregnancy (Women of child-bearing potential must have a negative pregnancy test prior to trial entry. Female patients of child-bearing potential and male patients with partners of child-bearing potential must agree to use adequate contraception methods, which must be continued for 3 months after completion of treatment
6. Patients with concurrent or previous malignancy that could compromise assessment of the primary and secondary endpoints of the trial; these cases must be discussed with UCL CTC prior to the patient being approached.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cohort 1 (limb soft tissue sarcomas): The rate of grade 2 or more late soft tissue fibrosis at 2 years following radiotherapy as assessed by RTOG late radiation morbidity criteria. | From date of registration until 2 years after date of registration.
  Late toxicity assessment measured using RTOG late radiation morbidity criteria.
Cohorts 2 (Ewing's sarcoma of the spine/pelvis): The proportion of patients in whom 90% of the planPTV receives 95% of the optimal prescription dose. | Upon completion of IMRT treatment
  Cohorts 2 (Ewing's sarcoma of the spine/pelvis): The proportion of patients in whom 90% of the planPTV receives 95% of the optimal prescription dose.
Cohort 3 (Non-Ewing's primary bone sarcomas of the spine/pelvis): The proportion of patients in whom 80% of the planPTV receives 95% of the optimal prescription dose. | Upon completion of IMRT treatment
  Cohort 3 (Non-Ewing's primary bone sarcomas of the spine/pelvis): The proportion of patients in whom 80% of the planPTV receives 95% of the optimal prescription dose.

SECONDARY OUTCOMES:
Acute RT toxicity - (For all cohorts) | From date of registration up to 90 days after date of registration
  In all 3 cohorts, Acute RT toxicity measured using RTOG acute radiation morbidity criteria.
Late RT toxicity - (For all cohorts) | From Day 91 after date of registration up to 3 years after date of registration
  In all 3 cohorts, late toxicities measured using the RTOG/EORTC Late Radiation Morbidity Scoring Criteria (skin, subcutaneous tissue fibrosis, bone, joint stiffness) and Stern's scale for oedema
Patient reported Quality of life (QOL) - (All cohorts) | Timepoints- Baseline, 1 year and 2 year post treatment
  All cohorts, patient reported Quality of life measured using EORTC QLQ-C30 quality of life questionnaire
Patient reported limb function (Cohort 1 only) | At timepoints - Baseline, 1 year and 2 years post Treatment
  For patients in Cohort 1 only, patient reported limb function measured using TESS questionnaire
Disease free survival (All Cohorts) | The start date for analysis will be the date of registration. From date of registration to date of documented disease progression assessed up to 3 years from date of registration
  Disease free survival will be calculated from the date of registration to date of documented disease progression, or death from any cause. Where progression is suspected and subsequently confirmed by scans, the date of documented suspected progression will be used. Patients alive and disease-free will be censored at the date last seen.
Overall survival (All Cohorts) | From date of registration to date of death or date of last follow-up assessment (assessed up to 3 years from date of registration)
  Overall survival time will be calculated from date of registration to the date of death from any cause or end of trial follow up
Time to local tumour recurrence (All Cohorts, for adjuvant RT) | From date of registration to date of documented recurrence within the irradiated site (assessed up to 3 years from date of registration)
  Time to local tumour recurrence evaluation from date of registration to first diagnosis of recurrence (histological or radiological).
Time to local disease progression (Cohorts 2 and 3, for definitive radical RT) | From date of registration to date of documented progression (assessed up to 3 years from date of registration)
  Time to local disease progression evaluation from date of registration to first diagnosis of progression.
Response by RECIST 1.1 (Cohorts 2 and 3, for definitive radical RT) | From date of registration to date of documented progression (assessed up to 3 years from date of registration)
  Response measured according to RECIST v 1.1 (for definitive radical RT)
Wound complications within 120 days of surgery (Cohort 1 only) | From date of definitive surgery until 120 days post surgery
  Rate and severity of wound complications assessed up to 120 days post surgery. This is a composite outcome measure assessed by a clinical examination of the wound.
For individual plans (cohort 2 & 3) | Upon completion of IMRT treatment.
  Percentage volume of planPTV receiving 95% of the prescription dose (50.4Gy/54Gy for cohort 2 and 60Gy/70Gy for cohort 3)
For individual plans (cohort 2 & 3) | Upon completion of IMRT treatment.
  Dose delivered to 95%, 80%, 70%, 60% and 50% volume of planPTV.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Seddon, Ph.D., M.D, Principal Investigator — University College London Hospitals
Locations (28):
- St Luke's Hospital, Dublin, Ireland
- United Kingdom (27):
  - Clatterbridge Cancer Centre, Bebington
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Adenbrookes' Hospital, Cambridge
  - Velindre Hospital, Cardiff
  - Cheltenham Hospital, Cheltenham
  - University Hospital Coventry, Coventry
  - Royal Derby Hospital, Derby
  - Western General Hospital, Edinburgh
  - Royal Devon & Exeter Foundation Trust, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James' Institute of Oncology, Leeds
  - Leicester Royal Infirmary, Leicester
  - University College London Hospitals, London
  - The Christie Hospital, Manchester
  - Northern Centre for Cancer Care, Newcastle
  - Northampton General Hospital, Northampton
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - The Royal Marsden NHS Foundation Trust, Sutton
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simoes R, Gulliford S, Seddon B, Dehbi HM, Robinson M, Forsyth S, Hughes A, Gaunt P, Nguyen TG, Elston S, Mohammed K, Zaidi S, Miles E, Hoskin P, Harrington K, Miah A. Predicting radiotherapy response, Toxicities and quality-of-life related functional outcomes in soft tissue sarcoma of the extremities (PredicT) using dose-volume constraints development: a study protocol. BMJ Open. 2024 Aug 9;14(8):e083617. doi: 10.1136/bmjopen-2023-083617. PMID 39122389
- [Derived] Simoes R, Miles E, Yang H, Le Grange F, Bhat R, Forsyth S, Seddon B. IMRiS phase II study of IMRT in limb sarcomas: Results of the pre-trial QA facility questionnaire and workshop. Radiography (Lond). 2020 Feb;26(1):71-75. doi: 10.1016/j.radi.2019.08.006. Epub 2019 Sep 14. PMID 31902458